## 1.5 OVERALL SYNOPSIS OF THE CLINICAL INVESTIGATION

| ANSM registration #: | 2022-A01183-40 |
|---|---|
| Clinical investigation plan #: | 22E0978 |
| Title of the clinical investigation: | SAFETY AND EFFECTIVENESS CLINICAL EVALUATION OF THE RANGE OF INJECTABLE MEDICAL DEVICES FILLGEL IN FACIAL AESTHETIC TREATMENT |
| Sponsor: | KYLANE LABORATOIRES SA Chemin du Pré-Fleuri 1-3 CH-1228 Plan-les-Ouates SWITZERLAND |
| Development phase | Exploratory study |
| Objectives: | The primary objective is to evaluate the effectiveness of the FILLGEL range used on different treated zones one month (M1) after treatment using clinical evaluation of the global aesthetic improvement (GAIS) rated by the independent investigator. The secondary objectives of the study are to collect data for the FILLGEL range on: |
| | <ul> <li>the effectiveness of the range used on different treated zones six months (M6) and twelve months (M12) after treatment using clinical evaluation of the global aesthetic improvement (GAIS) rated by the independent investigator.</li> <li>the safety using clinical evaluation of the Injection Site Reactions (ISR) rated by the subject and the investigator, and by collection of adverse events (AEs) at M1, M6 and M12.</li> <li>subject's satisfaction and subject's opinion on aesthetic improvement on the different treated zones using clinical evaluation of the GAIS at M1, M6 and M12.</li> <li>the injector's satisfaction on the injection quality using subjective evaluation questionnaire,</li> <li>Another objective will be to illustrate the device effectiveness by realization of face macrophotographs.</li> </ul> |
| Design: | <ul> <li>◆ Open study,</li> <li>◆ intra-individual,</li> <li>◆ single dose,</li> <li>◆ single centre.</li> </ul> |
| Planned Sample Size: | 68 subjects in total divided in 4 subgroups of 17 subjects, according to the kind of filler injected: Group 1: 17 subjects treated in peri-oral lines by FILLGEL 0 Group 2: 17 subjects treated in nasolabial folds and/or in lips by FILLGEL 1 (with at least 10 in nasolabial folds and 7 in lips, both indications possible on the same subjects). Group 3: 17 subjects treated in cheek/cheekbones by FILLGEL 2. Group 4: 17 subjects treated in cheek/cheekbones and/or chin by FILLGEL 3 (with at least 10 in cheeks/cheekbones and 7 in chin, both indications possible on the same subjects). |
| Number of investigational study sites: | 1 (Eurofins Dermscan Pharmascan) |

| KYLANE FILLGEL LABORATOIRES SA CIP #22E097 | Final version 2.0<br>Date: 21/09/2022 | Confidential<br>Page 13/74 |
|---|---|---|
|---|---|---|

| 2. Sex: male or female. 3. Age: between 18 and 65 years. 4. Subject seeking an improvement of her/his face aspect with HA filler. *For group_1: Subject with moderate to severe peri-oral lines (score 3 to 5 on Bazin Upper lip scale); *For group_2: Subject with moderate to severe nasolabial folds (score 3 to 4 on WSRS scale) and/or subject with his lips (score 1 or 2 for superior and/or inferior lip on the Rossi scale) and seeking an improvement of lip volume; *For group_3: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale); *For group_4: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale); *For group_4: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale) and/or subject seeking improvement of chin enhancement. 5. Subject whose weight did not fluctuate in the last 6 months and who agrees to keep a stable weight during the study. 6. Subject psychologically able to understand the information related to the study, and to give their written informed consent. 7. Subject psychologically able to understand the information related to the study, and to give their written informed consent. 8. Subject registered with a social security scheme. 9. Women of childbearing potential should use a contraceptive method considered effective since at least 4 weeks and throughout the study. Exclusion criteria: Exclusion criteria: Interms of population 1. Pregnant or nursing woman or planning a pregnancy during the study. 2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship. 3. Subject in a social or sanitary establishment. 4. Subject suspected to be non-compliant according to the investigator's judgment. 5. Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in research | | 1 Hoalthy Subject |
|---|---|---|
| 3. Age between 18 and 65 years. 4. Subject seeking an improvement of her/his face aspect with HA filler. *For group 1: Subject with moderate to severe peri-oral lines (score 3 to 5 on Bazin Upper lip scale); *For group 2: Subject with moderate to severe nasolabial folds (score 3 to 4 on WSRS scale) and/or subject with thin lips (score 1 or 2 for superior and/or inferior lip on the Rossi scale) and seeking an improvement of lip volume; *For group 3: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale); *For group 4: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale); *For group 4: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale) and/or subject seeking improvement of chin enhancement. 5. Subject whose weight did not fluctuate in the last 6 months and who agrees to keep a stable weight during the study. 6. Subject whose weight did not fluctuate in the last 6 months and who agrees to keep a stable weight during the study. 7. Subject having given their free, express, and informed consent. 8. Subject having given their free, express, and informed consent. 8. Subject having given their free, express, and informed consent. 9. Women of childbearing potential should use a contraceptive method considered effective since at least 4 weeks and throughout the study. 1. Pregnant or nursing woman or planning a pregnancy during the study. 2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship. 3. Subject suspected to be non-compliant according to the investigator's judgment. 4. Subject suspected to be non-compliant according to the investigator's judgment. 5. Subject winh and subject safety. 6. Subject with some history of suffering from autoimmune disease and/or immune deficiency. 8. Subject with some history of suffering from autoimmune disease and/or immune deficiency. 9. Subject with | Inclusion criteria: | Healthy Subject. Sex: male or female. |
| 4. Subject seeking an improvement of her/his face aspect with HA filler. *For. group. 1: Subject with moderate to severe peri-oral lines (score 3 to 5 on Bazin Upper lip scale); *For group 2: Subject with moderate to severe nasolabial folds (score 3 to 4 on WSRS scale) and/or subject with hin lips (score 1 or 2 for superior and/or inferior lip on the Rossi scale) and seeking an improvement of lip volume; *For group 3: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale); *For group 4: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale); *For group 4: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale) and/or subject seeking improvement of chin enhancement. 5. Subject whose weight did not fluctuate in the last 6 months and who agrees to keep a stable weight during the study. 6. Subject whose weight did not fluctuate in the last 6 months and who agrees to keep a stable weight during the study. 7. Subject psychologically able to understand then information related to the study, and to give their written informed consent. 8. Subject registered with a social security scheme. 9. Women of childbearing potential should use a contraceptive method considered effective since at least 4 weeks and throughout the study. Exclusion criteria: Exclusion criteria: Exclusion criteria: In terms of population 1. Pregnant or nursing woman or planning a pregnancy during the study. 2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship. 3. Subject in a social or sanitary establishment. 4. Subject who had been deprived of their preadomation in the study or whose non-enrollment period is not over. 5. Subject who had been deprived or their participation in research involving human beings in the last 12 months, including their participation in the present study. 6. Subject with sovan history of st | | |
| filler. *For group 1: Subject with moderate to severe peri-oral lines (score 3 to 5 on Bazin Upper lip scale); *For group 2: Subject with moderate to severe nasolabial folds (score 3 to 4 on WSRS scale) and/or subject with thin lips (score 1 or 2 for superior and/or inferior lip on the Rossi scale) and seeking an improvement of lip volume; *For group 3: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale); *For group 4: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale) and/or subject seeking improvement of chin enhancement. 5. Subject whose weight did not fluctuate in the last 6 months and who agrees to keep a stable weight during the study. 6. Subject having given their free, express, and informed consent. 7. Subject psychologically able to understand the information related to the study, and to give their written informed consent. 8. Subject having given their free, express, and informed consent. 8. Subject assistered with a social security scheme. 9. Women of childbearing potential should use a contraceptive method considered effective since at least 4 weeks and throughout the study. In terms of population 1. Pregnant or nursing woman or planning a pregnancy during the study. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship. 3. Subject in a social or sanitary establishment. 4. Subject suspected to be non-compliant according to the investigator's judgment. 5. Subject having received a total of 4,500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study. 6. Subject with sand/or subject safety. 6. Subject with sand/or subject safety. 9. Subject with some history of suffering from autoimmune disease and/or immune deficiency. 10. Subject with known history of suffering from autoimmune disease and/or immune deficiency. 1 | | |
| (score 3 to 5 on Bazin Upper lip scale); "For group_2 Subject with moderate to severe nasolabial folds (score 3 to 4 on WSRS scale) and/or subject with thin lips (score 1 or 2 for superior and/or inferior lip on the Rossi scale) and seeking an improvement of lip volume; "For group_3: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale); "For group_4: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale); "For group_4: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale) and/or subject seeking improvement of chin enhancement. Subject whose weight did not fluctuate in the last 6 months and who agrees to keep a stable weight during the study. Subject whose weight did not fluctuate in the last 6 months and who agrees to keep a stable weight during the study. Subject having given their free, express, and informed consent. Subject psychologically able to understand the information related to the study, and to give their written informed consent. Subject registered with a social security scheme. Women of childbearing potential should use a contraceptive method considered effective since at least 4 weeks and throughout the study. Interms of population 1. Pregnant or nursing woman or planning a pregnancy during the study. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship. 3. Subject in a social or sanitary establishment. 4. Subject suspected to be non-compliant according to the investigator's judgment. Subject is present study. Subject is uspected to be non-compliant according to the investigator's judgment. Subject is uspected to be non-compliant period is not over. Subject this free present study. Subject suspected to be non-compliant period is not over. Subject with known history of or suffering from autoimmune disease and/or is much estable. Interms of associated pathology | | filler. |
| For group 2: Subject with moderate to severe nasolabial folds (score 3 to 4 on WSRS scale) and/or subject with thin lips (score 1 or 2 for superior and/or inferior lip on the Rossi scale) and seeking an improvement of lip volume; | | |
| (score 3 to 4 on WSRS scale) and/or subject with thin lips (score 1 or 2 for superior and/or inferior lip on the Rossi scale) and seeking an improvement of lip volume; "For group 3: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale); "For group 4: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale) and/or subject seeking improvement of hin enhancement. Subject whose weight did not fluctuate in the last 6 months and who agrees to keep a stable weight during the study. Subject having given their free, express, and informed consent. Subject psychologically able to understand the information related to the study, and to give their written informed consent. Subject registered with a social security scheme. Women of childbearing potential should use a contraceptive method considered effective since at least 4 weeks and throughout the study. In terms of population 1. Pregnant or nursing woman or planning a pregnancy during the study. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship. Subject in a social or sanitary establishment. Subject suspected to be non-compliant according to the investigator's judgment. Subject suspected to be non-compliant according to the investigator's judgment. Subject suspected a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutane | | |
| i or 2 for superior and/or inferior lip on the Rossi scale) and seeking an improvement of lip volume; "For group 3: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale); "For group 4: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale) and/or subject seeking improvement of chin enhancement. 5. Subject whose weight did not fluctuate in the last 6 months and who agrees to keep a stable weight during the study. 6. Subject psychologically able to understand the information related to the study, and to give their written informed consent. 7. Subject psychologically able to understand the information related to the study, and to give their written informed consent. 8. Subject registered with a social security scheme. 9. Women of childbearing potential should use a contraceptive method considered effective since at least 4 weeks and throughout the study. 1. Pregnant or nursing woman or planning a pregnancy during the study. 2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship. 3. Subject in a social or sanitary establishment. 4. Subject suspected to be non-compliant according to the investigator's judgment. 5. Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study or whose non-enrollment period is not over. 7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject wiffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject wiffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disease and/or immun | | |
| seeking an improvement of lip volume; *For group 3: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale); *For group 4: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale) and/or subject seeking improvement of chin enhancement. 5. Subject whose weight did not fluctuate in the last 6 months and who agrees to keep a stable weight during the study. 6. Subject having given their free, express, and informed consent. 7. Subject psychologically able to understand the information related to the study, and to give their written informed consent. 8. Subject registered with a social security scheme. 9. Women of childbearing potential should use a contraceptive method considered effective since at least 4 weeks and throughout the study. 1. Pregnant or nursing woman or planning a pregnancy during the study. 2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship. 3. Subject in a social or sanitary establishment. 4. Subject suspected to be non-compliant according to the investigator's judgment. 5. Subject having received a total of 4.500 euros as compensations for their participation in research inviting human beings in the last 12 months, including their participation in the present study. 6. Subject enrolled in another study or whose non-enrollment period is not over. 7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosaceae, porphyria) in the 6 months before screening visit. 1. Subject with | | |
| "For group 3: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale); "For group 4: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale); "For group 4: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale) and/or subject seeking improvement of chin enhancement. 5. Subject whose weight did not fluctuate in the last 6 months and who agrees to keep a stable weight during the study. 6. Subject having given their free, express, and informed consent. 7. Subject psychologically able to understand the information related to the study, and to give their written informed consent. 8. Subject registered with a social security scheme. 9. Women of childbearing potential should use a contraceptive method considered effective since at least 4 weeks and throughout the study. In terms of population 1. Pregnant or nursing woman or planning a pregnancy during the study. 2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship. 3. Subject in a social or sanitary establishment. 4. Subject suspected to be non-compliant according to the investigator's judgment. 5. Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study. 6. Subject enrolled in another study or whose non-enrollment period is not over. 7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disease and | | |
| Ilipoatrophy scale : "For group 4: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale) and/or subject seeking improvement of chin enhancement. | | · |
| *For group 4: Subject with moderate to severe cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale) and/or subject seeking improvement of chin enhancement. 5. Subject whose weight did not fluctuate in the last 6 months and who agrees to keep a stable weight during the study. 6. Subject having given their free, express, and informed consent. 7. Subject psychologically able to understand the information related to the study, and to give their written informed consent. 8. Subject registered with a social security scheme. 9. Women of childbearing potential should use a contraceptive method considered effective since at least 4 weeks and throughout the study. Exclusion criteria: In terms of population 1. Pregnant or nursing woman or planning a pregnancy during the study. 2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship. 3. Subject in a social or sanitary establishment. 4. Subject suspected to be non-compliant according to the investigator's judgment. 5. Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study. 6. Subject enrolled in another study or whose non-enrollment period is not over. 7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency. 10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit. | | |
| cheeks/cheekbones volume deficit (score 3 to 4 on Ascher lipoatrophy scale) and/or subject seeking improvement of chin enhancement. 5. Subject whose weight did not fluctuate in the last 6 months and who agrees to keep a stable weight during the study. 6. Subject having given their free, express, and informed consent. 7. Subject psychologically able to understand the information related to the study, and to give their written informed consent. 8. Subject registered with a social security scheme. 9. Women of childbearing potential should use a contraceptive method considered effective since at least 4 weeks and throughout the study. In terms of population 1. Pregnant or nursing woman or planning a pregnancy during the study. 2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship. 3. Subject in a social or sanitary establishment. 4. Subject suspected to be non-compliant according to the investigator's judgment. 5. Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study. 6. Subject enrolled in another study or whose non-enrollment period is not over. 7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency. 10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit. 11. Subject with a history of streptococcal disease or an active streptococcus infection. | | |
| lipoatrophy scale) and/or subject seeking improvement of chin enhancement. 5. Subject whose weight did not fluctuate in the last 6 months and who agrees to keep a stable weight during the study. 6. Subject having given their free, express, and informed consent. 7. Subject psychologically able to understand the information related to the study, and to give their written informed consent. 8. Subject registered with a social security scheme. 9. Women of childbearing potential should use a contraceptive method considered effective since at least 4 weeks and throughout the study. Exclusion criteria: In terms of population 1. Pregnant or nursing woman or planning a pregnancy during the study. 2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship. 3. Subject in a social or sanitary establishment. 4. Subject suspected to be non-compliant according to the investigator's judgment. 5. Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study. 6. Subject enrolled in another study or whose non-enrollment period is not over. 7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit. 11. Subject with ha history of streptococcal disease or an active streptococcus infection. | | |
| enhancement. 5. Subject whose weight did not fluctuate in the last 6 months and who agrees to keep a stable weight during the study. 6. Subject having given their free, express, and informed consent. 7. Subject psychologically able to understand the information related to the study, and to give their written informed consent. 8. Subject registered with a social security scheme. 9. Women of childbearing potential should use a contraceptive method considered effective since at least 4 weeks and throughout the study. Interms of population 1. Pregnant or nursing woman or planning a pregnancy during the study. 2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship. 3. Subject in a social or sanitary establishment. 4. Subject suspected to be non-compliant according to the investigator's judgment. 5. Subject having received a total of 4,500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study. 6. Subject enrolled in another study or whose non-enrollment period is not over. 7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency. 10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit. 11. Subject with a history of streptococcal disease or an active streptococcus infection. | | |
| 5. Subject whose weight did not fluctuate in the last 6 months and who agrees to keep a stable weight during the study. 6. Subject having given their free, express, and informed consent. 7. Subject psychologically able to understand the information related to the study, and to give their written informed consent. 8. Subject registered with a social security scheme. 9. Women of childbearing potential should use a contraceptive method considered effective since at least 4 weeks and throughout the study. Exclusion criteria: In terms of population 1. Pregnant or nursing woman or planning a pregnancy during the study. 2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship. 3. Subject in a social or sanitary establishment. 4. Subject suspected to be non-compliant according to the investigator's judgment. 5. Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study. 6. Subject enrolled in another study or whose non-enrollment period is not over. 7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency. 10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit. 11. Subject with a history of streptococcal disease or an active streptococcus infection. | | |
| who agrees to keep a stable weight during the study. 6. Subject having given their free, express, and informed consent. 7. Subject psychologically able to understand the information related to the study, and to give their written informed consent. 8. Subject registered with a social security scheme. 9. Women of childbearing potential should use a contraceptive method considered effective since at least 4 weeks and throughout the study. Interms of population 1. Pregnant or nursing woman or planning a pregnancy during the study. 2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship. 3. Subject in a social or sanitary establishment. 4. Subject suspected to be non-compliant according to the investigator's judgment. 5. Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study. 6. Subject enrolled in another study or whose non-enrollment period is not over. 7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency. 10. Subject suffering from a stive disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screeni | | |
| 7. Subject psychologically able to understand the information related to the study, and to give their written informed consent. 8. Subject registered with a social security scheme. 9. Women of childbearing potential should use a contraceptive method considered effective since at least 4 weeks and throughout the study. In terms of population 1. Pregnant or nursing woman or planning a pregnancy during the study. 2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship. 3. Subject in a social or sanitary establishment. 4. Subject suspected to be non-compliant according to the investigator's judgment. 5. Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study. 6. Subject enrolled in another study or whose non-enrollment period is not over. 7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency. 10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit. 11. Subject with a history of streptococcal disease or an active streptococcus infection. | | |
| related to the study, and to give their written informed consent. 8. Subject registered with a social security scheme. 9. Women of childbearing potential should use a contraceptive method considered effective since at least 4 weeks and throughout the study. In terms of population 1. Pregnant or nursing woman or planning a pregnancy during the study. 2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship. 3. Subject in a social or sanitary establishment. 4. Subject suspected to be non-compliant according to the investigator's judgment. 5. Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study. 6. Subject enrolled in another study or whose non-enrollment period is not over. 7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency. 10. Subject with known history and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit. 11. Subject with a history of streptococcal disease or an active streptococcus infection. | | |
| 8. Subject registered with a social security scheme. 9. Women of childbearing potential should use a contraceptive method considered effective since at least 4 weeks and throughout the study. In terms of population 1. Pregnant or nursing woman or planning a pregnancy during the study. 2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship. 3. Subject in a social or sanitary establishment. 4. Subject suspected to be non-compliant according to the investigator's judgment. 5. Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study. 6. Subject enrolled in another study or whose non-enrollment period is not over. 7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency. 10. Subject wiffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit. 11. Subject with a history of streptococcal disease or an active streptococcus infection. | | |
| 9. Women of childbearing potential should use a contraceptive method considered effective since at least 4 weeks and throughout the study. In terms of population 1. Pregnant or nursing woman or planning a pregnancy during the study. 2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship. 3. Subject in a social or sanitary establishment. 4. Subject suspected to be non-compliant according to the investigator's judgment. 5. Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study. 6. Subject enrolled in another study or whose non-enrollment period is not over. 7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency. 10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit. 11. Subject with a history of streptococcal disease or an active streptococcus infection. | | |
| Exclusion criteria: In terms of population | | |
| throughout the study. In terms of population 1. Pregnant or nursing woman or planning a pregnancy during the study. 2. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship. 3. Subject in a social or sanitary establishment. 4. Subject suspected to be non-compliant according to the investigator's judgment. 5. Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study. 6. Subject enrolled in another study or whose non-enrollment period is not over. 7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency. 10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit. 11. Subject with a history of streptococcal disease or an active streptococcus infection. | | |
| Exclusion criteria: In terms of population | | |
| <ol> <li>Pregnant or nursing woman or planning a pregnancy during the study.</li> <li>Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.</li> <li>Subject in a social or sanitary establishment.</li> <li>Subject suspected to be non-compliant according to the investigator's judgment.</li> <li>Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study.</li> <li>Subject enrolled in another study or whose non-enrollment period is not over.</li> <li>Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up).</li> <li>In terms of associated pathology</li> <li>Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety.</li> <li>Subject with known history of or suffering from autoimmune disease and/or immune deficiency.</li> <li>Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit.</li> <li>Subject with a history of streptococcal disease or an active streptococcus infection.</li> </ol> | Exclusion criteria: | |
| <ol> <li>Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.</li> <li>Subject in a social or sanitary establishment.</li> <li>Subject suspected to be non-compliant according to the investigator's judgment.</li> <li>Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study.</li> <li>Subject enrolled in another study or whose non-enrollment period is not over.</li> <li>Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up).</li> <li>In terms of associated pathology</li> <li>Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety.</li> <li>Subject with known history of or suffering from autoimmune disease and/or immune deficiency.</li> <li>Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit.</li> <li>Subject with a history of streptococcal disease or an active streptococcus infection.</li> </ol> | | |
| administrative or legal decision or who is under guardianship. 3. Subject in a social or sanitary establishment. 4. Subject suspected to be non-compliant according to the investigator's judgment. 5. Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study. 6. Subject enrolled in another study or whose non-enrollment period is not over. 7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency. 10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit. 11. Subject with a history of streptococcal disease or an active streptococcus infection. | | |
| guardianship. 3. Subject in a social or sanitary establishment. 4. Subject suspected to be non-compliant according to the investigator's judgment. 5. Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study. 6. Subject enrolled in another study or whose non-enrollment period is not over. 7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency. 10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit. 11. Subject with a history of streptococcal disease or an active streptococcus infection. | | |
| <ol> <li>Subject in a social or sanitary establishment.</li> <li>Subject suspected to be non-compliant according to the investigator's judgment.</li> <li>Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study.</li> <li>Subject enrolled in another study or whose non-enrollment period is not over.</li> <li>Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up).</li> <li>In terms of associated pathology</li> <li>Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety.</li> <li>Subject with known history of or suffering from autoimmune disease and/or immune deficiency.</li> <li>Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit.</li> <li>Subject with a history of streptococcal disease or an active streptococcus infection.</li> </ol> | | |
| <ol> <li>Subject suspected to be non-compliant according to the investigator's judgment.</li> <li>Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study.</li> <li>Subject enrolled in another study or whose non-enrollment period is not over.</li> <li>Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up).</li> <li>In terms of associated pathology</li> <li>Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety.</li> <li>Subject with known history of or suffering from autoimmune disease and/or immune deficiency.</li> <li>Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit.</li> <li>Subject with a history of streptococcal disease or an active streptococcus infection.</li> </ol> | | |
| <ol> <li>Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study.</li> <li>Subject enrolled in another study or whose non-enrollment period is not over.</li> <li>Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up).</li> <li>In terms of associated pathology</li> <li>Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety.</li> <li>Subject with known history of or suffering from autoimmune disease and/or immune deficiency.</li> <li>Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit.</li> <li>Subject with a history of streptococcal disease or an active streptococcus infection.</li> </ol> | | |
| compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study. 6. Subject enrolled in another study or whose non-enrollment period is not over. 7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency. 10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit. 11. Subject with a history of streptococcal disease or an active streptococcus infection. | | |
| human beings in the last 12 months, including their participation in the present study. 6. Subject enrolled in another study or whose non-enrollment period is not over. 7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency. 10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit. 11. Subject with a history of streptococcal disease or an active streptococcus infection. | | |
| participation in the present study. 6. Subject enrolled in another study or whose non-enrollment period is not over. 7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency. 10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit. 11. Subject with a history of streptococcal disease or an active streptococcus infection. | | |
| <ol> <li>Subject enrolled in another study or whose non-enrollment period is not over.</li> <li>Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up).</li> <li>In terms of associated pathology <ol> <li>Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety.</li> <li>Subject with known history of or suffering from autoimmune disease and/or immune deficiency.</li> </ol> </li> <li>Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit.</li> <li>Subject with a history of streptococcal disease or an active streptococcus infection.</li> </ol> | | |
| period is not over. 7. Subject with scar(s), mole(s), hair or any other lesion on the studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency. 10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit. 11. Subject with a history of streptococcal disease or an active streptococcus infection. | | |
| studied zones which might interfere with the evaluation (tattoo, permanent make-up). In terms of associated pathology 8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety. 9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency. 10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit. 11. Subject with a history of streptococcal disease or an active streptococcus infection. | | |
| <ul> <li>(tattoo, permanent make-up).</li> <li>In terms of associated pathology</li> <li>8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety.</li> <li>9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency.</li> <li>10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit.</li> <li>11. Subject with a history of streptococcal disease or an active streptococcus infection.</li> </ul> | | |
| <ul> <li>In terms of associated pathology</li> <li>8. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety.</li> <li>9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency.</li> <li>10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit.</li> <li>11. Subject with a history of streptococcal disease or an active streptococcus infection.</li> </ul> | | |
| <ol> <li>Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety.</li> <li>Subject with known history of or suffering from autoimmune disease and/or immune deficiency.</li> <li>Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit.</li> <li>Subject with a history of streptococcal disease or an active streptococcus infection.</li> </ol> | | (tattoo, permanent make-up). |
| <ol> <li>Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results and/or subject safety.</li> <li>Subject with known history of or suffering from autoimmune disease and/or immune deficiency.</li> <li>Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit.</li> <li>Subject with a history of streptococcal disease or an active streptococcus infection.</li> </ol> | | In terms of associated pathology |
| <ul> <li>any other pathology that may interfere with the evaluation of the study results and/or subject safety.</li> <li>9. Subject with known history of or suffering from autoimmune disease and/or immune deficiency.</li> <li>10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit.</li> <li>11. Subject with a history of streptococcal disease or an active streptococcus infection.</li> </ul> | | |
| <ol> <li>Subject with known history of or suffering from autoimmune disease and/or immune deficiency.</li> <li>Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit.</li> <li>Subject with a history of streptococcal disease or an active streptococcus infection.</li> </ol> | | |
| disease and/or immune deficiency. 10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit. 11. Subject with a history of streptococcal disease or an active streptococcus infection. | | the study results and/or subject safety. |
| <ul> <li>10. Subject suffering from active disease such as inflammation, infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit.</li> <li>11. Subject with a history of streptococcal disease or an active streptococcus infection.</li> </ul> | | |
| infection, tumours, inflammatory and/or infectious cutaneous disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit. 11. Subject with a history of streptococcal disease or an active streptococcus infection. | | |
| disorders (herpes, acne, rosacea, porphyria) in the 6 months before screening visit. 11. Subject with a history of streptococcal disease or an active streptococcus infection. | | |
| months before screening visit. 11. Subject with a history of streptococcal disease or an active streptococcus infection. | | |
| 11. Subject with a history of streptococcal disease or an active streptococcus infection. | | |
| streptococcus infection. | | |
| · | | |
| 12. Oubject profite to develop illimations skill conditions of | | 12. Subject prone to develop inflammatory skin conditions or |
| having tendency to bleeding disorders. | | |

| 🛟 eurofins | Dermscan | PRM03-F-227_V6_EN |
|------------|------------|--------------------------------------|
| | Pharmascan | Clinical investigational plan for MD |

| KYLANE<br>LABORATOIRES SA | FILLGEL<br>CIP #22E0978 | Final version 2.0<br>Date: 21/09/2022 | Confidential<br>Page 14/74 |
|---|---|---|---|
| LABORATORIZOGA | 13. Sub hav 14. Sub sho ingranti ana trea 15. Sub hya Relating to 16. Any the 17. Sub or r che derr plar 18. Sub plar of th (e.g mes zon 19. Sub perr Poly 20. Sub inflathro inje 22. Sub | pject predisposed to keloids ing healing disorders. Dject having history of several ck including known hyperedients of the investigation (Diasept esthetics (EMLA®), related the testhetics of the testhetics of the testhetics (EMLA®), related the testhetics of the testhetic | or hypertrophic scarring of the sensitivity to one of the onal device (i.e. HA), to onal device or current ersensitivity reactions to one of the onal device of the coverage of the onal derivation. Interpretation of the onal derivation of the onal derivation of the past 6 months or who one of the past 18 months of the |
| | mor<br>24. Sub<br>stud<br>25. Sub | nsive exposure to sunlight or<br>onth and/or planning to do so<br>opject planning to change he | during the study. er/his life habits during the esumption of alcohol (more |

| Investigational device: |
|-------------------------|
| Name / code |

Galenic form Indication

FILLGEL range: Injectable sterile gels in syringe

1. FILLGEL 0: Indication: Peri-oral lines

2. FILLGEL 1: Indication: Nasolabial folds / lip volume

3. FILLGEL 2: Indication: Cheeks, cheekbones

| KYLANE | FILLGEL | Final version 2.0 | Confidential |
|-----------------|--------------|-------------------|--------------|
| LABORATOIRES SA | CIP #22E0978 | Date: 21/09/2022 | Page 15/74 |

| LABORATOIRES SA | CIP #22E0978 | P #22E0978 Date: 21/09/2022 Page 15/74 | |
|---|---|---|---|
| | 4. FILL GEL | . 3: Indication: Cheeks, chee | ekbones / chin |
| Endpoints: | Primary end | | <u> </u> |
| Lindpoints. | Proportion of with the ovindependen An improvei | Proportion of subjects having an improvement of the zone treated with the overall FILLGEL range of devices as assessed by the independent investigator, one month after treatment, using the GAIS. An improvement is defined as a subject with "very much improved", "much improved" or "improved" score on the GAIS. | |
| | Secondary 6 | endpoints: | |
| | - The safet | • | nd of each FILLGEL device |
| | (ISI | | arly Injection Site Reactions aily-log every day up to one |
| | inve<br>mo | | arly ISRs by the independent one (M1), six (M6) and twelve e study. |
| | with the ov | rerall FILLGEL range of d<br>t investigator, six and twe | rovement of the zone treated evices as assessed by the elve months after treatment, |
| | with each F assessed b | ILLGEL device for the four | rovement of the zone treated indications independently as igator, one, six and twelve |
| | with the FI | LLGEL range of devices | rovement of the zone treated overall as assessed by the ter treatment, using the GAIS. |
| | with each F assessed by | ILLGEL device for the four | rovement of the zone treated indications independently as , and twelve months after |
| | FILLGEL 0 independen | used in the peri-oral | nkles/lines filling of the device<br>lines as assessed by the<br>welve months after treatment,<br>e. |
| | 1 used in t | the nasolabial folds as as one, six and twelve month | s filling of the device FILLGEL sessed by the independent as after treatment, using the |
| | FILLGEL 1 i | | volume increase of the device<br>the independent investigator<br>nent, using the Rossi scale. |

| eurofins | Dermscan |
|----------|------------|
| | Pharmascan |

- Evaluation of the effectiveness on volume restauration of the device FILLGEL 2 used in the cheeks/cheekbones as assessed by the

independent investigator, one, six and twelve months after treatment, using the Ascher lipoatrophy scale.

| KYLANE<br>LABORATOIRES SA | LGEL Final version 2.0 Confidential 22E0978 Date: 21/09/2022 Page 16/74 | | |
|---|---|---|---|
| | - Evaluation of the effectiveness on volume restauration of the device FILLGEL 3 used in the cheeks/cheekbones as assessed by the independent investigator, one, six and twelve months after treatment, using the Ascher lipoatrophy scale. | | |
| | | atisfaction on the injection<br>nmediately after injection o | quality using a questionnaire<br>n D0. |
| | | of the treatment effect one mpared to baseline by pho | , six and twelve months after tographs taking. |
| Study Procedures: | Screening, D | 0, D7 (phone call for safety | y), M1, M6, M12 |
| Statistical methods: | The statistica | I analysis will be performe | d by the CRO biostatistician. |
| | on the ITT ar<br>The analysis<br>performed or | nd PP population.<br>s of the secondary effect<br>n the ITT and PP populati | e parameter will be performed<br>viveness parameters will be<br>ion. In case the ITT and PP<br>ily the PP population will be |
| | The analysis<br>the "safety" p | | ameters will be performed on |
| | A descriptive analysis of the population will be performed, including subject's characteristics, subject's disposition, deviations to the protocol, injections characteristics. | | |
| | For the primary evaluation criteria: | | |
| | For the parameter GAIS investigator with the <u>5 level scores</u> (at D0 after injection, M1, M6 and M12), the frequencies and percentages will be presented for the <b>overall face score</b> and for the scores <b>by product</b> . | | |
| | Two derived parameters will be defined based on the parameters GAIS subject and investigator as a scores of 2 levels (1=Improvement (Very much improved, Much improved and Improved) and 2=No change or worsening). At each time point, these parameters will be described in frequencies, percentages and Confidence Interval (CI) 95%. | | |
| | Inferential a | nalysis for the primary ev | valuation criteria |
| | For the new derived parameters at M1 (1 month after injection) for the GAIS Investigator, a binomial exact test (bilateral approach) vs 50% will be applied at each time point for the <b>overall face score</b> . This test will compare the proportion of improvement to 50%. | | |
| | For the secondary evaluation criteria: | | <u>ı:</u> |
| | All the variables will be described using adapted statistics according to their type (quantitative data or qualitative data). Statistical tests will be performed, to assess the change from baseline (Wilcoxon signed rank test). | | |
| | The bilateral | approach will be used with | a significance level of 0.05. |

| KYLANE | FILLGEL | Final version 2.0 | Confidential |
|-----------------|--------------|-------------------|--------------|
| LABORATOIRES SA | CIP #22E0978 | Date: 21/09/2022 | Page 17/74 |
| LADORATOIREO DA | | | 9 |

| Estimated dates of the study: | Clinical investigation beginning: Q4 2022 |
|---|---|
| | Clinical investigation end: Q4 2023/Q1 2024 |
| | Expected recruitment period duration: 3 months |
| | Clinical investigation overall duration: 12 months + recruitment period |
| | Duration by subject: 12 months + screening period |

KYLANE FILLGEL Final version 2.0 Confidential LABORATOIRES SA CIP #22E0978 Date: 21/09/2022 Page 18/74

## **FLOW-CHART**

| LOW-CHART | | | | | | |
|---|---|---|---|---|---|---|
| Procedure | Visit 1<br>Screening | Visit 2<br>Day 0 | Phone call<br>Day 7 | Visit 3<br>M1 | Visit 4<br>M6 | Visit 5<br>M12 |
| Days | D-x | D0 | D7 ± 1 | D30±7 | D180±14 | D365±14 |
| Informed consent form signature | • | | | | | |
| Medical examination | • | | | | | |
| Medical history and previous and concomitant treatments collection | • | | | | | |
| Verification of the inclusion and exclusion criteria | • | | | | | |
| Urinary pregnancy test (for women with childbearing potential) | | <b>●</b> b | | | | |
| Confirmation of eligibility | | ● <sup>b</sup> | | | | |
| Photographs (full face + 2 profiles) | | ●p | | • | • | • |
| Scoring of effectiveness using specific scales | | ● b | | • | • | • |
| Injection | | • | | | | |
| Injector satisfaction questionnaire | | <b>⊕</b> a | | | | |
| GAIS live assessment by the independent investigator | | ea | | • | • | • |
| GAIS assessment by the subjects | | | | • | • | • |
| Distribution of a subject daily-log | • | • | | • | • | • |
| ISR collection by subject | Each day during one month after injection, on the daily-log | | | | | |
| ISR investigator | | ● <sup>a</sup> | | • | • | • |
| AE and concomitant treatments and procedures collection | • | • | • | • | • | • |

a : after injection, b : before injection

AE: Adverse Event - GAIS: Global Aesthetic Improvement Scale- ISR: Injection Site Reaction